CLINICAL TRIAL: NCT05723731
Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Chronic Constipation: A Randomized Controlled Trial
Brief Title: Effect of Transcutaneous Auricular Vagal Nerve Stimulation on Chronic Constipation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A pre-specified interim analysis was conducted as planned, we calculated a P-value greater than 0.57 when comparing response rates between taVNS and sham group, resulting in an early termination of the study.
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20222075-F-1
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Chronic Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation | interventions — Laxatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): patients will receive taVNS at left tragus for four weeks.
  Interventions: Device: taVNS; Drug: Laxative Agent
- Sham-treatment group (Sham Comparator): patients will receive sham-taVNS at left earlobe for four weeks.
  Interventions: Device: taVNS; Drug: Laxative Agent

INTERVENTIONS:
Device: taVNS — Patients will receive taVNS (device produced by Xi'an Bashui Health Technology Co., Ltd) thirty minutes twice a day in the morning and the night for four weeks (duty circle: 30s "on" periods and 30s "off" periods; frequency: 25 Hz; amplitude of 0-2 mA at the maximum level that the patient could tolerate; pulse width: 0.5ms)
Drug: Laxative Agent — Bisacodyl or glycerin enemas can be used in patients who do not have a bowel movement for more than 3 days.

SUMMARY:
The worldwide prevalence of chronic constipation (CC) is 15%, and women are more likely to develop the disease than men. CC have a significant impact on quality of life and increase the burden of national health insurance. The conventional medication treatments are primarily symptom-specific and have limited efficacy. Previous small sample study had shown the therapeutic potential of transcutaneous auricular vagus nerve stimulation (taVNS) for irritable bowel syndrome with constipation (IBS-C). The aim of this study was to investigate whether taVNS could improve defecation condition and constipation symptoms in patients with CC.

ELIGIBILITY:
Inclusion Criteria:

1. FC or IBS-C patients aged 18-75 years who meet the diagnostic criteria for Rome IV;
2. Complete spontaneous bowel movements (CSBMs) per week < 3;
3. No constipation medication used for at least 2 weeks prior to enrollment, not participated in clinical trials in the past three months, and no abnormal colonoscopy within the past 12 months in those with alarm symptoms.

Exclusion Criteria:

1. Have cognitive impairment, psychiatric disorders, or conditions that may affect patient cooperation;
2. Have a cardiac pacemaker implantation or other electronically implanted devices;
3. Prior taVNS treatment;
4. History of colorectal surgery, except for simple appendectomy;
5. Severe cardiovascular, hepatic, or renal disease;
6. Known malignancy;
7. Secondary constipation caused by medications and other diseases;
8. Pregnant or lactating women;
9. Refusal to sign an informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Responder rate | 4 weeks
  Proportion of patients with an average of 3 or more complete spontaneous bowel movements (CSBMs) per week from 1 to 4 weeks

SECONDARY OUTCOMES:
Responder rate at the time of the follow-up visit | 8 weeks
  Proportion of patients with an average of 3 or more CSBMs per week from 5 to 12 weeks
CSBMs | 12 weeks
  Changes from baseline by time point in the CSBMs
Spontaneous bowel movements (SBMs) | 12 weeks
  Changes from baseline by time point in the SBMs
Abdominal symptoms | 12 weeks
  Changes from baseline by time point in abdominal symptoms scores (abdominal bloating, abdominal fullness, abdominal discomfort, abdominal pain, abdominal cramping).
Bristol stool form scale (BFSF) | 12 weeks
  Changes from baseline by time point in the BFSF
Laxative agents using | 12 weeks
  Proportion of patients using laxative agents and/or other adjunctive bowel measures at 1-12 weeks and the average number of times per week
Patient Assessment of Constipation symptom (PAC-SYM) | 12 weeks
  Changes from baseline by time point in the PAC-SYM score
Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL) | 12 weeks
  Changes from baseline by time point in the PAC-QOL score
Self-Rating Depression Scale (SDS) | 12 weeks
  Changes from baseline by time point in SDS scores
Self-Rating Anxiety Scale (SAS) | 12 weeks
  Changes from baseline by time point in SAS scores
Adverse events | 12 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Department of Gastroenterology, Second Affiliated Hospital, Lanzhou University, Lanzhou, Gansu
  - Department of Gastroenterology, National Clinical Research Center of Infectious Disease, The Third People's Hospital of Shenzhen, The Second Affiliated Hospital of Southern University of Science and Technology, Shenzhen, Guangdong
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Xijing 986 Hospita, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact PI to get IPD.

REFERENCES:
- [Result] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Result] Nag A, Martin SA, Mladsi D, Olayinka-Amao O, Purser M, Vekaria RM. The Humanistic and Economic Burden of Chronic Idiopathic Constipation in the USA: A Systematic Literature Review. Clin Exp Gastroenterol. 2020 Jul 16;13:255-265. doi: 10.2147/CEG.S239205. eCollection 2020. PMID 32765039
- [Result] Shi X, Hu Y, Zhang B, Li W, Chen JD, Liu F. Ameliorating effects and mechanisms of transcutaneous auricular vagal nerve stimulation on abdominal pain and constipation. JCI Insight. 2021 Jul 22;6(14):e150052. doi: 10.1172/jci.insight.150052. PMID 34138761
- [Derived] Liu T, Wang Z, Li Y, Kang X, Wang X, Ren G, Lv Y, Li J, Liu Y, Liang S, Wang X, Huang X, Zhang X, Wang J, Nie Y, Luo H, Sun J, Qin W, Han Y, Pan Y. Effects of Transcutaneous Auricular Vagal Nerve Stimulation on Chronic Constipation: A Multicenter, Randomized Controlled Study. United European Gastroenterol J. 2025 Oct;13(8):1550-1559. doi: 10.1002/ueg2.70041. Epub 2025 May 13. PMID 40359320